CLINICAL TRIAL: NCT06105294
Title: Time-Restricted Eating as an Adjunctive Intervention for Bipolar Disorder: Acceptability and Feasibility
Brief Title: Time-Restricted Eating and Bipolar Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decided to shift to a new design and measures
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-10-15725
Record Dates: First submitted 2023-02-06; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Bipolar Disorder
Keywords: eating; circadian
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Participants will take part in a baseline assessment, then all will be assigned to time-restricted eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- time-restricted eating (Experimental): Post-baseline, participants will be asked to restrict their eating to a 10-hour window.
  Interventions: Behavioral: time-restricted eating

INTERVENTIONS:
Behavioral: time-restricted eating — Restrict eating to a 10-hour window.

SUMMARY:
This is a pilot trial to examine the acceptability and feasibility of time-restricted eating as an adjunct to medication treatment for bipolar disorder.

DETAILED DESCRIPTION:
Time-restricted eating (TRE) is a way of scheduling food intake that has been shown to improve circadian rhythms in animals and humans. TRE is based on animal and human science that shows that the timing of eating powerfully influences diurnal rhythms. Animal research has shown that feeding during sleep periods leads to a surge of norepinephrine, cortisol, wakefulness, and activity. Drawing on this, over a decade of studies have examined the impact of experimentally randomizing mice to time-restricted feeding during wake hours (vs. 24-hour ad libitum feeding). Importantly, caloric intake and other facets of diet were yoked for strict control. A consistent finding is that TRE had powerful benefits for circadian and metabolic indicators across studies,and more recent data also shows benefit for animal longevity.

Here, the investigators' goal is to extend this work to bipolar disorder (BD). More specifically, the investigators will gather data to examine the acceptability and feasibility of TRE among those who self-identify with bipolar disorder and who experience some problems with sleep, circadian rhythms, or schedules. The investigators will gather measures of mania, depression, sleep, and QOL, to provide preliminary evidence of change on these dimensions.

ELIGIBILITY:
Inclusion Criteria:

* adults diagnosed with bipolar disorder and currently receiving medical care for their bipolar disorder.
* Experiencing schedule/sleep or circadian problem in the past 3 months
* Medication regimens stable for past month
* Adequate English language skills for taking part in the program.
* Living in California.

Exclusion Criteria:

* Cognitive deficits (Screening OMC Test)
* Current: psychosis, (hypo)mania, major depressive episode, substance/alcohol use disorders, eating disorder diagnoses or acute suicidal risk (MINI interview; see DSM5 TRE screening)
* High scores (> 5) on the Screening Eating Disorder Examination Questionnaire
* Current shift work
* >5 kg weight change within 3 months
* Pregnancy
* Breastfeeding
* Uncorrected hypo or hyperthyroidism

  * diabetes type 1
* Gastrointestinal conditions impairing nutrient absorption
* Medications contraindicated for fasting, including clozapine, glucose-lowering medications, diabetes-related injections, requiring food early morning or late evening, corticosteroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Acceptability as assessed using self-ratings on items designed for this study | Immediately post-treatment (10 weeks)
  self-ratings of the acceptability of the intervention
Feasibility as assessed by percent of clients who complete the assessments and intervention | Immediately post-treatment (10 weeks)
  Percentage of clients who do not drop out of the trial. Drop out would be defined as not completing the TRE intervention, or failing to complete the end-of-treatment intervention.

SECONDARY OUTCOMES:
Lower Mania symptoms as assessed with the Patient Mania Questionnaire-9 | Change from baseline to immediately post-treatment (10 weeks)
  Self-Rated Patient Mania Questionnaire-9
Lower Depression symptoms as assessed with the Patient Health Questionnaire-9 | Change from baseline to immediately post-treatment (10 weeks)
  PHQ-9
Lower scores on two Patient Reported Outcome Measurement Information System (PROMIS) sleep scales | Change from baseline to immediately post-treatment (10 weeks)
  PROMIS self-report of sleep disturbance and sleep-related impairment (summed together)
higher scores on Self-rated Quality of Life | Change from baseline to immediatly post-treatment (10 weeks)
  Brief Quality of Life in Bipolar Disorder scale

OTHER OUTCOMES:
Higher Functional impairment on the World Health Organization Disability Assessment Schedule (WHO-DAS2.0) | Change from baseline to immediatly post-treatment (10 weeks)
  WHO-DAS2.0 nonphysical health-related scales

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available at OSF post-study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of study completion, if ethics board approves.
Access Criteria: Available through OSF.

REFERENCES:
- See also: link to study team website — https://calm.berkeley.edu/participate/